CLINICAL TRIAL: NCT03158155
Title: Prevalence of Early Childhood Caries in Egyptian Children With Serum Vitamin D Deficiency.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nancy Ahmed El Salmawy (Other)
Responsible Party: Sponsor-Investigator, Nancy Ahmed El Salmawy, Principal Investigator,, Cairo University
Organization: Cairo University (Other)
Other Study IDs: CEBD-2017-5-101
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood samples will be obtained from children recruited in the study at the day of diagnosis, seven mm of blood will collect approximately, using radioimmunoassay technique for measuring vitamin D serum level All serum analysis will be done in Radioisotope Department, Nuclear Research Center, and Atomic Energy Authority.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with vitamin D deficiency: 1. children with vitamin D deficiency with age group from 2-5 years old

SUMMARY:
To detect the effect of vitamin D deficiency in the development of early childhood caries (ECC) among Egyptian children.

DETAILED DESCRIPTION:
Justification for undertaking the trial:

American Academy of Pediatric Dentistry (2012), defined early childhood caries (ECC) as the presence of one or more decayed, missing teeth (resulting from caries), or filled surfaces in the primary tooth of child 6 years old or younger.

Early childhood caries is a chronic childhood disease, that decreasing quality of life, this include pain, disturbed sleep, poor aesthetics, difficulty in eating and speaking and behavioral changes that affect the child's self-esteem. (Guay, 2004).

Due to the rising incidence of dental carries in early childhood, contributory factors need to be investigated in order to facilitate treatment of such a large population of children in desperate need of dental care (Guay, 2004).These multiple risk factors include the lack of a dental home, poor oral hygiene, diet, and nutrition ( Najeeb et al., 2016).

Enamel is the most mineralized substance in the human body; it is mainly made of calcium and phosphate. Vitamin D plays an important role in increasing the absorption of calcium and phosphate from food. Which calcium and phosphate improve the strength of the teeth as make them able to fight the demineralization from bacteria (Youssef et al., 2011). Therefore, it is responsible of promoting the calcification of teeth, having a topical fluoride like effect, and in the forming of enamel, dentin, and bone. (Mellanby & Pattison, 1928).

Vitamin D receptors are present on the cells of immune system and on the teeth. It binds to these receptors and increases the amount of good antimicrobial proteins as cathelicidin and other special defense in saliva (Youssef et al., 2011). These antimicrobial peptides have antibacterial neutralizing activity against periodonto pathogens as gram negative and gram positive bacteria and candida albicans, its effective in vitro against oral microorganisms such as streptococcus mutants, prophyromonas gingivalis and actinobacillus, so it prevents dental caries.( Potturu et al., 2014).

East, (1939) study concluded that children who consumed a high vitamin D diet, vitamin D played an indispensable role in 1) preventing the initiation of new caries, 2) inhibiting the spread of existing caries, and 3) arresting the caries. Likewise, an examination of children found a decreased caries prevalence in areas of increased vitamin D exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages from two to five years
2. Both sexes.
3. Parent and children cooperation.
4. Healthy children.
5. Children with serum vitamin D deficiency.

Exclusion Criteria:

1. Children age more than 5 years.
2. Children had a complex metabolic or medical disorder.
3. Parents that will not sign the consent.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Egyptain children age ranges from 2 to 5 years from Abo El Rish Hospital, Malnutrition clinic.
Sampling Method: Probability Sample
Enrollment: 288 (Estimated)
Dates: Start 2017-07-15 (Estimated); Primary Completion 2018-07-15 (Estimated); Study Completion 2018-07-18 (Estimated)

PRIMARY OUTCOMES:
Prevalence of early childhood caries | 6 months
  Stages of Early childhood caries.
  1. Initial (reversible stage)
  2. Damaged (carious) stage
  3. Deep lesions
  4. Traumatic stage.
  5. Arrested caries.

SECONDARY OUTCOMES:
Delayed tooth formation and eruption | 6 months
  * Delayed tooth eruption.
  * Tooth smaller than normal
Gingivitis | 6 months
  binary yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Nourhan A. El dokky, A. Professor, Study Director — neldokky@hotmail.com

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Policy on Early Childhood Caries (ECC): Classifications, Consequences, and Preventive Strategies. Pediatr Dent. 2016 Oct;38(6):52-54. No abstract available. PMID 27931420
- [Background] Anthonappa, R. P., and King, N. M. (2015). Enamel defects in the permanent dentition: prevalence and etiology. Springer-Verlag Berlin Heidelberg 2015; B.K. Drummond, N. Kilpatrick (eds.), Planning and Care for Children and Adolescents with Dental Enamel Defects: Etiology, Research and Contemporary Management, pp. 15-30
- [Background] Antonenko O, Bryk G, Brito G, Pellegrini G, Zeni SN. Oral health in young women having a low calcium and vitamin D nutritional status. Clin Oral Investig. 2015 Jul;19(6):1199-206. doi: 10.1007/s00784-014-1343-x. Epub 2014 Oct 31. PMID 25359326
- [Background] Baumann, F., Jäger, E., & Bloch, W. (2013).Vitamin D -office of dietary supplements-National instituted health. Journal of Molecular Modeling
- [Background] Bener, A., Al Darwish, M. S., and Hoffmann , G. F. (2013). Vitamin D deficiency and risk of dental caries among young children: A public health problem. Indian Journal of Oral Sciences, 4(2): 75-82
- [Background] Bener A, Alsaied A, Al-Ali M, Al-Kubaisi A, Basha B, Abraham A, Guiter G, Mian M. High prevalence of vitamin D deficiency in type 1 diabetes mellitus and healthy children. Acta Diabetol. 2009 Sep;46(3):183-9. doi: 10.1007/s00592-008-0071-6. Epub 2008 Oct 10. PMID 18846317
- [Background] Wagner CL, Greer FR; American Academy of Pediatrics Section on Breastfeeding; American Academy of Pediatrics Committee on Nutrition. Prevention of rickets and vitamin D deficiency in infants, children, and adolescents. Pediatrics. 2008 Nov;122(5):1142-52. doi: 10.1542/peds.2008-1862. PMID 18977996
- [Background] Douglass JM, Douglass AB, Silk HJ. A practical guide to infant oral health. Am Fam Physician. 2004 Dec 1;70(11):2113-20. PMID 15606059
- [Background] Dudding T, Thomas SJ, Duncan K, Lawlor DA, Timpson NJ. Re-Examining the Association between Vitamin D and Childhood Caries. PLoS One. 2015 Dec 21;10(12):e0143769. doi: 10.1371/journal.pone.0143769. eCollection 2015. PMID 26692013
- [Background] East BR. Mean Annual Hours of Sunshine and the Incidence of Dental Caries. Am J Public Health Nations Health. 1939 Jul;29(7):777-80. doi: 10.2105/ajph.29.7.777. No abstract available. PMID 18015076
- [Background] Fuleihan Gel-H, Bouillon R, Clarke B, Chakhtoura M, Cooper C, McClung M, Singh RJ. Serum 25-Hydroxyvitamin D Levels: Variability, Knowledge Gaps, and the Concept of a Desirable Range. J Bone Miner Res. 2015 Jul;30(7):1119-33. doi: 10.1002/jbmr.2536. Epub 2015 May 7. PMID 25952470
- [Background] Grant WB. A review of the role of solar ultraviolet-B irradiance and vitamin D in reducing risk of dental caries. Dermatoendocrinol. 2011 Jul;3(3):193-8. doi: 10.4161/derm.3.3.15841. Epub 2011 Jul 1. PMID 22110779
- [Background] Guay AH. Access to dental care: solving the problem for underserved populations. J Am Dent Assoc. 2004 Nov;135(11):1599-605; quiz 1623. doi: 10.14219/jada.archive.2004.0088. PMID 15622666
- [Background] Herzog K, Scott JM, Hujoel P, Seminario AL. Association of vitamin D and dental caries in children: Findings from the National Health and Nutrition Examination Survey, 2005-2006. J Am Dent Assoc. 2016 Jun;147(6):413-20. doi: 10.1016/j.adaj.2015.12.013. Epub 2016 Jan 27. PMID 26827077
- [Background] Krall EA, Wehler C, Garcia RI, Harris SS, Dawson-Hughes B. Calcium and vitamin D supplements reduce tooth loss in the elderly. Am J Med. 2001 Oct 15;111(6):452-6. doi: 10.1016/s0002-9343(01)00899-3. PMID 11690570
- [Background] Mellanby M, Pattison CL. THE ACTION OF VITAMIN D IN PREVENTING THE SPREAD AND PROMOTING THE ARREST OF CARIES IN CHILDREN. Br Med J. 1928 Dec 15;2(3545):1079-82. doi: 10.1136/bmj.2.3545.1079. No abstract available. PMID 20774325
- [Background] Najeeb S, Zafar MS, Khurshid Z, Zohaib S, Almas K. The Role of Nutrition in Periodontal Health: An Update. Nutrients. 2016 Aug 30;8(9):530. doi: 10.3390/nu8090530. PMID 27589794
- [Background] Youssef DA, Miller CW, El-Abbassi AM, Cutchins DC, Cutchins C, Grant WB, Peiris AN. Antimicrobial implications of vitamin D. Dermatoendocrinol. 2011 Oct;3(4):220-9. doi: 10.4161/derm.3.4.15027. Epub 2011 Oct 1. PMID 22259647
- [Background] Potturu, M., Prabhakaran, P. A., Oommen, N., Sarojini, D. M., and Sunil, S. N.(2014). Cathelicidin expression and role in oral health and diseases: A short review. Tropical J. of Med. Res., 17 (2): 69-75.
- [Background] Schroth RJ, Lavelle C, Tate R, Bruce S, Billings RJ, Moffatt ME. Prenatal vitamin D and dental caries in infants. Pediatrics. 2014 May;133(5):e1277-84. doi: 10.1542/peds.2013-2215. PMID 24753535
- [Result] American Academy of Pediatric Dentistry Clinical Affairs Committee; American Academy of Pediatric Dentistry Council on Clinical Affairs. Guideline on periodicity of examination, preventive dental services, anticipatory guidance, and oral treatment for children. Pediatr Dent. 2005-2006;27(7 Suppl):84-6. No abstract available. PMID 16541901